CLINICAL TRIAL: NCT02127437
Title: Lanreotide In Polycystic Kidney Disease Study
Acronym: LIPS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: IPSEN pharmaceutical company, Boulogne-Billancourt, France (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LIPS-01
Record Dates: First submitted 2014-04-02; First posted 2014-04-30 (Estimated); Last update posted 2019-11-18 (Actual); Status verified 2019-11

CONDITIONS: Autosomal Dominant Polycystic Kidney Disease (ADPKD
Keywords: Autosomal dominant polycystic kidney disease,; Glomerular filtration rate,; Somatostatin,; lanreotide
MeSH Terms: conditions — Polycystic Kidney, Autosomal Dominant | interventions — lanreotide; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A - treated group (Experimental)
  Interventions: Drug: Lanreotide
- B - control group (Placebo Comparator)
  Interventions: Drug: saline

INTERVENTIONS:
Drug: Lanreotide — 120 mg, subcutaneously, once every 4 weeks
  Arms: A - treated group
Drug: saline — 0,5 ml, subcutaneously, once every 4 weeks
  Arms: B - control group

SUMMARY:
LIPS study (Lanreotide In Polycystic kidney disease Study) is a prospective randomized double blind placebo controlled study. The main objective is to prove that lanreotide, a somatostatin analog, is able to reduce the glomerular filtration rate decline over 3 years by at least 30%. Cardiovascular outcomes, blood pressure, quality of life and safety are among the secondary outcomes. The study, which will include 180 ADPKD patients, is scheduled to start in early 2014.

An equal number of patients with chronic kidney disease stage 2 (90 patients with GFR 89 to 60 ml/mn/1.73 m2) and chronic kidney disease stage 3 (90 patients with GFR 59 to 30 ml/mn/1.73 m2) will be included. The primary endpoint (GFR decline) will be assessed by repeated measures, in the overall population as well as in the two GFR stratus.

ELIGIBILITY:
Inclusion Criteria:

* autosomal dominant polycystic kidney disease (clinical, familial, imaging grounds)
* measured GFR : 30 to 89 ml/mn/1.73m2
* age > 18
* affiliated with health insurance
* written informed consent

Exclusion Criteria:

* iohexol /iodine allergy
* diabetes mellitus
* other associated nephropathy suspected
* evolutive or recent malignant disease ( in the previous 5 years)
* cholelithiasis
* uncontrolled hypertension (BP>160/100 mmHg)
* cardiac failure of grade III or IV according to the NYHA (New York Heart Association) classification
* liver failure
* psychiatric illness
* pregnancy, lactation, lack of contraception
* use of somatostatin analogs during the last 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 159 (Actual)
Dates: Start 2014-09-19 (Actual); Primary Completion 2019-07-31 (Actual); Study Completion 2019-07-31 (Actual)

PRIMARY OUTCOMES:
Glomerular filtration rate (GFR) | month 36

SECONDARY OUTCOMES:
Glomerular filtration rate (GFR) | month 18
Glomerular filtration rate (GFR) decline | month 36
Safety, tolerance | month 36
Onset or worsening of hypertension | month 18
Onset or worsening of hypertension | month 36
Quality of life | month 0
  SF-36, EQ5D
Quality of life | month 18
  SF-36, EQ5D
Quality of life | month 36
  SF-36, EQ5D
Cystic pain | month 36

CONTACTS AND LOCATIONS:
Overall Officials: Dominique JOLY, MD, PhD, Principal Investigator — Necker hospital
Locations (1):
- Necker hospital, Paris, France

REFERENCES:
- [Derived] St Pierre K, Cashmore BA, Bolignano D, Zoccali C, Ruospo M, Craig JC, Strippoli GF, Mallett AJ, Green SC, Tunnicliffe DJ. Interventions for preventing the progression of autosomal dominant polycystic kidney disease. Cochrane Database Syst Rev. 2024 Oct 2;10(10):CD010294. doi: 10.1002/14651858.CD010294.pub3. PMID 39356039